CLINICAL TRIAL: NCT06165458
Title: Clinical Comparison of Whitening Efficacy and Tooth Sensitivity of Different Concentrations of Hydrogen Peroxide Photoactivated With Violet or Blue LEDs
Brief Title: Whitening Efficacy and Tooth Sensitivity of Different Concentrations of Hydrogen Peroxide Photoactivated With Violet or Blue LEDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: UFPara017
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Color; Bleaching Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HP6V (Experimental): 6% hydrogen peroxide gel + violet LED
  Interventions: Other: 6% hydrogen peroxide gel + violet LED
- HP6B (Experimental): 6% hydrogen peroxide gel + blue LED
  Interventions: Other: 6% hydrogen peroxide gel + blue LED
- HP35V (Experimental): 35% hydrogen peroxide gel + violet LED
  Interventions: Other: 35% hydrogen peroxide gel + violet LED
- HP35B (Experimental): 35% hydrogen peroxide gel + blue LED
  Interventions: Other: 35% hydrogen peroxide gel + blue LED

INTERVENTIONS:
Other: 6% hydrogen peroxide gel + violet LED — Tooth whitening with 6% hydrogen peroxide gel (Lase Peroxide Lite, DMC, São Carlos, Brazil) activated by violet LED
  Arms: HP6V
Other: 6% hydrogen peroxide gel + blue LED — Tooth whitening with 6% hydrogen peroxide gel (Lase Peroxide Lite, DMC, São Carlos, Brazil) activated by blue LED
  Arms: HP6B
Other: 35% hydrogen peroxide gel + violet LED — Tooth whitening with 35% hydrogen peroxide gel (Lase Peroxide Sensy, DMC, São Carlos, Brazil) activated by violet LED
  Arms: HP35V
Other: 35% hydrogen peroxide gel + blue LED — Tooth whitening with 35% hydrogen peroxide gel (Lase Peroxide Sensy, DMC, São Carlos, Brazil) activated by blue LED
  Arms: HP35B

SUMMARY:
This is a randomized, controlled, double-blind and repeated-measures clinical trial evaluated the photoactivation of hydrogen peroxide gels in different concentrations with blue or violet LED in terms of whitening efficacy and tooth sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* at age 18 or older, with good general and oral health;
* possessing all six natural and healthy upper anterior teeth with a color shade of A2 or darker, determined by comparison with the Vita Classic scale;

Exclusion Criteria:

* pregnant and breastfeeding women;
* individuals with internal tooth discoloration (tetracycline stains, fluorosis or hypoplasias);
* smokers, or those with veneers or restorations on the teeth in questions were excluded;
* gingival recession;
* dentin exposure;
* periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Color | Color assessment was carried out before bleaching, 1 week after bleaching and 3 months after bleaching
  A operator measured the color of the six upper anterior teeth using a digital spectrophotometer (VITA Easyshade V, Wilcos, Petrópolis, RJ, Brazil).
Bleaching Sensitivity | Assessments were carried out three times: before bleaching, immediately after bleaching, and 24 hours after bleaching.
  The degree of tooth sensitivity of patients was recorded using a visual analogue scale (VAS) from 0 to 10, where 0 represents no tooth sensitivity and 10 represents the greatest tooth sensitivity ever felt by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pará, Belém, Pará, Brazil

REFERENCES:
- [Derived] Oliveira MGVV, Dutra DJB, Costa JLSG, Besegato JF, Barros APO, Oliveira RR, Araujo PV, Alvim HH. Clinical comparison of whitening efficacy and tooth sensitivity of different concentrations of hydrogen peroxide photoactivated with violet or blue LEDs. Lasers Med Sci. 2024 Jul 26;39(1):195. doi: 10.1007/s10103-024-04144-6. PMID 39060473